CLINICAL TRIAL: NCT06506370
Title: Nonsurgical Periodontal Care for Diabetes Patients: A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Arturo Sánchez-Pérez, Profesor Contratado Doctor Permanente, Universidad de Murcia
Other Study IDs: ID: 141/2013, March 3, 2013
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis; Diabetes
Keywords: periodontitis; glycosylated haemoglobin; glycaemic control; nonsurgical periodontal therapy; periodontal disease
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients without periodontitis and with diabetes.: Periodontitis was diagnosed in patients who presented with attachment losses due to inflammatory problems greater than or equal to 2 mm at the interproximal level or greater than or equal to 3 mm at the buccal or lingual/palatal level in two or more nonadjacent teeth.
  The diagnosis of diabetes was made at the endocrinology service of the Hospital Virgen de la Arrixaca in Murcia.
  Interventions: Other: nonsurgical periodontal treatment
- Test group: Patients with periodontitis and diabetes.: Periodontitis was diagnosed in patients who presented with attachment losses due to inflammatory problems greater than or equal to 2 mm at the interproximal level or greater than or equal to 3 mm at the buccal or lingual/palatal level in two or more nonadjacent teeth.
  The diagnosis of diabetes was made at the endocrinology service of the Hospital Virgen de la Arrixaca in Murcia.
  Interventions: Other: nonsurgical periodontal treatment

INTERVENTIONS:
Other: nonsurgical periodontal treatment — The patients underwent treatment in accordance with the guidelines of the European Federation of Periodontology (EFP). Initially, patients were informed of their condition, educated on oral hygiene practices, and advised to cease detrimental habits such as smoking. Following this, supragingival cleaning was conducted using ultrasound, with manual subgingival instrumentation utilizing a reduced set of Gracey curettes for pockets exceeding 4 mm with persistent bleeding or greater than 6 mm.

SUMMARY:
Diabetes mellitus (DM) and periodontitis are two chronic diseases that are interconnected. The coexistence of these conditions leads to increased severity of periodontitis and challenges in controlling blood glucose levels in diabetic patients. The aim of the present study was to evaluate both the influence of periodontal disease and its treatment in patients with DM in terms of a reduction in glycosylated haemoglobin levels at 3 and 6 months after treatment.

DETAILED DESCRIPTION:
A sequential, nonprobabilistic, controlled, prospective and longitudinal case-control study was carried out at the University Dental Clinic of the Morales Meseguer Hospital in Murcia, Spain. Thirty diabetic patients were divided into two groups. Participants were assigned to either the periodontal treatment group (test group), which received oral hygiene instructions along with scaling and root planing utilizing ultrasound and Gracey curettes, or the nonperiodontal group (control group), which received oral hygiene instructions along with supragingival removal of plaque and calculus using ultrasound. Periodontal and endocrine-metabolic variables were evaluated at baseline and at 3 and 6 months. Clinical periodontal variables such as the plaque index (PI), bleeding on probing (BOP), periodontal probing depth (PPD), clinical attachment level (CAL), and glycosylated haemoglobin (HbA1c) levels were assessed.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included individuals who met the following specifications: diagnosed with diabetes mellitus, aged 18 years or older, exhibited moderate or advanced periodontitis (clinical insertion loss of 2 mm interproximally or exceeding 3 mm vestibularly or linguodistally in more than 2 nonadjacent teeth), and possessed an HbA1c level between 5.5 and 11. Additionally, participants were allowed to participate in the study only if they did not have any significant diabetic complications and completed the informed consent forms indicating their willingness to participate in the present study.

Exclusion Criteria:

* The exclusion criteria were as follows: patients previously diagnosed and treated for periodontal disease; pregnant or lactating patients; individuals who had taken antibiotics, antiseptics, or medications that could affect the host response during the month prior to the periodontal assessment; patients with uncontrolled DM; and patients who did not sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty diabetic patients (15 periodontal and 15 nonperiodontal patients; 8 women and 22 men; 5 smokers and 25 nonsmokers) with a mean age of 55 years were included in the present study. The mean duration of diabetes was 19 years. The patients were referred by the endocrinology service of the Virgen de la Arrixaca University Hospital in Murcia (Spain) to the University Dental Clinic of the Morales Meseguer Hospital in Murcia (Spain) for periodontal clinical examination by the same trained person (B.M-M.).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Level of glycosylated haemoglobin (HbA1c) | All the samples were reviewed at 3 and 6 months after treatment, and all the periodontal and endocrine-metabolic variables mentioned above were noted.
  The HbA1c test is expressed as a percentage, with a normal range being below 5.7%, prediabetes between 5.7% and 6.4%, and diabetes 6.5% or higher.

SECONDARY OUTCOMES:
Plaque index | All the samples were reviewed at 3 and 6 months after treatment, and all the periodontal and endocrine-metabolic variables mentioned above were noted.
  The plaque index is a clinical measure used to assess the amount of dental plaque on teeth. It evaluates the thickness and extent of plaque accumulation on the tooth surfaces. Typically, a scoring system is used, ranging from 0 (no plaque) to 3 (abundant plaque)
Bleeding on probing | All the samples were reviewed at 3 and 6 months after treatment, and all the periodontal and endocrine-metabolic variables mentioned above were noted.
  Bleeding on probing (BOP) is a clinical sign used in dentistry to assess gum health. It occurs when gentle probing of the gums around the teeth causes bleeding, indicating inflammation or infection, such as gingivitis or periodontitis.
Periodontal probing depth | All the samples were reviewed at 3 and 6 months after treatment, and all the periodontal and endocrine-metabolic variables mentioned above were noted.
  Periodontal probing depth is the measurement of the space between the gum and the tooth, from the top of the gumline to the bottom of the pocket. This is done using a periodontal probe and is used to assess the health of the gums and diagnose periodontal disease. Healthy gums typically have probing depths of 1-3 mm.
Clinical attachment level | All the samples were reviewed at 3 and 6 months after treatment, and all the periodontal and endocrine-metabolic variables mentioned above were noted.
  Clinical attachment level (CAL) is the measurement from the cementoenamel junction (CEJ) to the base of the periodontal pocket. It indicates the extent of periodontal support loss around a tooth, combining probing depth and gum recession. CAL is crucial for diagnosing and monitoring periodontal disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Odontológica Universitaria, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data of the present study are available as Excel files upon request to the corresponding author (arturosa@um.es).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Indefined